CLINICAL TRIAL: NCT00000593
Title: Viral Activation Transfusion Study (VATS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 313
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2005-12

CONDITIONS: Acquired Immunodeficiency Syndrome; Blood Transfusion; Cytomegalovirus Infections; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cytomegalovirus Infections; HIV Infections | interventions — Blood Transfusion

INTERVENTIONS:
Procedure: blood transfusion

SUMMARY:
The purpose of the trial was to determine if transfusion of allogeneic blood to HIV-1 infected persons led to immune activation and consequent induction of HIV-1 or /or Cytomegalovirus (CMV) replication, and whether this adversely affected clinical prognosis.

DETAILED DESCRIPTION:
BACKGROUND:

The initiative was approved by the NHLBI AIDS Ad Hoc Working Group and given concept clearance by the September 1993 National Heart, Lung, and Blood Advisory Council. The initiative was released in January 1994.

DESIGN NARRATIVE:

Patient enrollment started in August 1995. Patients scheduled for transfusion were entered into the study at the time of their first transfusion and randomized to receive leukopoor red cells filtered within 24 hours of collection or unmanipulated blood components. Patients received blood as per their treatment arm as needed for one or two years. Patients were stratified to those with CD4 counts below 50 /MM3 (most patients) and those with CD4 counts above that level. Primary endpoints were overall survival and a change in HIV viremia after the 1st transfusion. The secondary endpoint was the occurrence of a new AIDS-defining complication. A substudy looked at donor lymphocytes in the immunosuppressed recipients to help determine why AIDS patients don't seem to get post-transfusion graft-vs-host disease. The patient recruitment time was extended for one year because of low accrual. With new drugs, especially protease inhibitors, the proportion of patients needing transfusion has decreased. The patients are less severely ill and their disease produces less anemia. Furthermore, the new drugs don't have anemia as a side effect. The trial ended in January, 2000.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
HIV-infected patients with CD4 counts below 250 who clinically needed red blood cell transfusions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-11; Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Kalish — New England Research Institute, Inc.

REFERENCES:
- [Background] Busch MP, Collier A, Gernsheimer T, Carrington JD, Flanigan TP, Kashkari M, Kennedy M, Kumar PN, Lane TA, Mellors JW, Mohandas K, Pollard RB, Viele M, Yomtovian R, Holland PV, McCurdy PR. The Viral Activation Transfusion Study (VATS): rationale, objectives, and design overview. Transfusion. 1996 Oct;36(10):854-9. doi: 10.1046/j.1537-2995.1996.361097017169.x. No abstract available. PMID 8863770
- [Background] Lee TH, Sakahara NS, Fiebig EW, Hirschkorn DF, Johnson DK, Busch MP. Quantitation of white cell subpopulations by polymerase chain reaction using frozen whole-blood samples. Viral Activation Transfusion Study. Transfusion. 1998 Mar;38(3):262-70. doi: 10.1046/j.1537-2995.1998.38398222870.x. PMID 9563406
- [Background] Kalish LA, Collier AC, Flanigan TP, Kumar PN. Plasma human immunodeficiency virus (HIV) type 1 RNA load in men and women with advanced HIV-1 disease. J Infect Dis. 2000 Aug;182(2):603-6. doi: 10.1086/315710. Epub 2000 Jul 21. PMID 10915096
- [Background] Collier AC, Kalish LA, Busch MP, Gernsheimer T, Assmann SF, Lane TA, Asmuth DM, Lederman MM, Murphy EL, Kumar P, Kelley M, Flanigan TP, McMahon DK, Sacks HS, Kennedy MS, Holland PV; Viral Activation Transfusion Study Group. Leukocyte-reduced red blood cell transfusions in patients with anemia and human immunodeficiency virus infection: the Viral Activation Transfusion Study: a randomized controlled trial. JAMA. 2001 Mar 28;285(12):1592-601. doi: 10.1001/jama.285.12.1592. PMID 11268267
- [Background] Lane TA, Gernsheimer T, Mohandas K, Assmann SF. Signs and symptoms associated with the transfusion of WBC-reduced RBCs and non-WBC-reduced RBCs in patients with anemia and HIV infection: results from the Viral Activation Transfusion Study. Transfusion. 2002 Feb;42(2):265-74. doi: 10.1046/j.1537-2995.2002.00036.x. PMID 11896345
- [Background] Brecher ME, Triulzi DJ, Assmann SF; Viral Activation Transfusion Study. Number of RBC units and rate of transfusionto anemic HIV-positive patients assigned to receiveWBC-reduced or non-WBC-reduced RBCs: the viral activation transfusion study experience. Transfusion. 2001 Jun;41(6):794-8. doi: 10.1046/j.1537-2995.2001.41060794.x. PMID 11399822
- [Background] Kennedy MS, Kalish LA, Mohandas K, Gernsheimer T, Townsend-McCall D; Viral Activation Transfusion Study Group. The transfusion trigger and number of units transfused in patients with HIV: associations with disease stage and functional status. Transfusion. 2002 Apr;42(4):456-61. doi: 10.1046/j.1525-1438.2002.00081.x. PMID 12076293
- [Background] Asmuth DM, Kalish LA, Laycock ME, Murphy EL, Mohr BA, Lee TH, Gallarda J, Giachetti C, Dollard SC, van der Horst CM, Grant RM, Busch MP; Viral Activation Transfusion Study Group. Absence of HBV and HCV, HTLV-I and -II, and human herpes virus-8 activation after allogeneic RBC transfusion in patients with advanced HIV-1 infection. Transfusion. 2003 Apr;43(4):451-8. doi: 10.1046/j.1537-2995.2003.00350.x. PMID 12662277
- [Background] Ariga H, Lee TH, Laycock ME, Mohr BA, Kalish LA, Yomtovian R, Gernsheimer T, Busch MP; Viral Activation Transfusion Study. Residual WBC subsets in filtered prestorage RBCs. Transfusion. 2003 Jan;43(1):98-106. doi: 10.1046/j.1537-2995.2003.00270.x. PMID 12519437
- [Background] Drew WL, Chou S, Miner RC, Mohr BA, Busch MP, van der Horst CM, Asmuth DM, Kalish LA. Cytomegalovirus glycoprotein B groups in human immunodeficiency virus-infected patients with incident retinitis. J Infect Dis. 2002 Jul 1;186(1):114-7. doi: 10.1086/341071. Epub 2002 May 22. PMID 12089671
- [Background] Eisenbud R, Assmann SF, Kalish LA, van Der Horst C, Collier AC; Viral Activation Transfusion Study Group. Differences in difficulty adjudicating clinical events in patients with advanced HIV disease. J Acquir Immune Defic Syndr. 2001 Sep 1;28(1):43-6. doi: 10.1097/00042560-200109010-00007. PMID 11579276
- [Background] Yomtovian R, Gernsheimer T, Assmann SF, Mohandas K, Lee TH, Kalish LA, Busch MP; Viral Activation Transfusion Study Group. WBC reduction in RBC concentrates by prestorage filtration: multicenter experience. Transfusion. 2001 Aug;41(8):1030-6. doi: 10.1046/j.1537-2995.2001.41081030.x. PMID 11493735
- [Background] Kruskall MS, Lee TH, Assmann SF, Laycock M, Kalish LA, Lederman MM, Busch MP; Viral Activation Transfusion Study Group. Survival of transfused donor white blood cells in HIV-infected recipients. Blood. 2001 Jul 15;98(2):272-9. doi: 10.1182/blood.v98.2.272. PMID 11435293
- [Background] Murphy EL, Collier AC, Kalish LA, Assmann SF, Para MF, Flanigan TP, Kumar PN, Mintz L, Wallach FR, Nemo GJ; Viral Activation Transfusion Study Investigators. Highly active antiretroviral therapy decreases mortality and morbidity in patients with advanced HIV disease. Ann Intern Med. 2001 Jul 3;135(1):17-26. doi: 10.7326/0003-4819-135-1-200107030-00005. PMID 11434728
- [Background] Para MF, Kalish LA, Collier AC, Murphy EL, Drew WL; Viral Activation Transfusion Study Group. Correlates of change in cytomegalovirus viremia in patients with advanced human immunodeficiency virus infection who require transfusion. J Infect Dis. 2001 Jun 1;183(11):1673-7. doi: 10.1086/320702. Epub 2001 Apr 27. PMID 11343218
- [Background] Para MF, Kalish LA, Collier AC, Pollard RB, Kumar PN, Mintz L, Wallach FR, Drew WL; Viral Activation Transfusion Study (VATS) Group. Qualitative and quantitative PCR measures of cytomegalovirus in patients with advanced HIV infection who require transfusions. J Acquir Immune Defic Syndr. 2001 Apr 1;26(4):320-5. doi: 10.1097/00126334-200104010-00004. PMID 11317072
- Available data/document: Individual Participant Data Set: VATS — http://biolincc.nhlbi.nih.gov/studies/vats/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/vats/